CLINICAL TRIAL: NCT01266863
Title: E Test Strips Applied to Bronchoalveolar Lavage for Suspicion of Hospital-acquired Pneumonia to Accelerate Antibiogram Analysis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Victor Segalen Bordeaux 2 (Other)
Responsible Party: Principal Investigator, Alexandre Boyer, Medical doctor, Université Victor Segalen Bordeaux 2
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ABoyer3
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Hospital-acquired Pneumonia
Keywords: Hospital-acquired pneumonia; E test; Antibiogram; Bronchoalveolar lavage
MeSH Terms: conditions — Healthcare-Associated Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- E test method (Experimental)
  Interventions: Other: E test method

INTERVENTIONS:
Other: E test method — E test strips directly applied to BAL

SUMMARY:
To rapidly adapt or deescalate the initially broad antibiotic treatment, an antibiogram analysis is required. E test strips have successfully provided an antibiogram 24 h after having been directly applied to bronchoalveolar lavage (BAL). An open-label, prospective cohort study of consecutive patients with hospital-acquired pneumonia will be conducted with the aim of validating a new method increasing the rapidity of antibiogram analysis compared to standard methods of culture. This antibiogram will be provided by E test strips directly applied to bronchoalveolar lavage (BAL) samples and analyzed from the 6th up to the 24th hour after its completion. The occurrence of major errors (S with E test method, I or R with standard method) and minor errors (I or R with E test method and S with standard method)will be observed and a comparison of H6, H10 and H24 results performed.

ELIGIBILITY:
Inclusion Criteria:

* all patients with suspected HAP undergoing BAL will be eligible

Exclusion Criteria:

* contraindications for BAL (PaO2/FIO2 <100, risk of bronchoscopy-related haemorrhagic complications), secondary exclusion of patients with negative cultures, defined by a threshold of bacteria <104 CFU/ml.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Major error defined as the MIC(s) classified as R or I by E test method and S by referent method | 2 days

SECONDARY OUTCOMES:
Minor error defined as the MIC(s) classified as R or I by E test method and S by referent method | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

REFERENCES:
- [Derived] Boyer A, Goret J, Clouzeau B, Romen A, Prevel R, Lhomme E, Vargas F, Hilbert G, Bebear C, Gruson D, M'Zali F. Tailoring Empirical Antimicrobial Therapy in Subjects With Ventilator-Associated Pneumonia With a 10-Hour E-Test Approach. Respir Care. 2019 Mar;64(3):307-312. doi: 10.4187/respcare.06255. Epub 2018 Dec 11. PMID 30538161